CLINICAL TRIAL: NCT05902455
Title: Differential Mobility Spectrometry (DMS) Based Oral Tumor Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Olfactomics Oy (Unknown)
Responsible Party: Sponsor
Other Study IDs: R20100L(a)
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-06

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Oral squamous cell carcinoma; Differential mobility spectrometry (DMS); Automatic tissue analysis (ATAS)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — * Punch biopsy (4mm) of oral squamous cell carcinoma tumor
  * Control biopsy (4mm) of healthy oral mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with oral squamous cell carcinoma
  Interventions: Procedure: Punch biopsy

INTERVENTIONS:
Procedure: Punch biopsy — Punch biopsy of oral squamous cell carcinoma tumor and a control biopsy of healthy oral mucosa are collected during primary tumor excision surgery from each recruited patient.

SUMMARY:
The trial is a single-center, non-randomized feasibility study aiming to evaluate the feasibility of ex-vivo tissue analysis using differential mobility spectrometry (DMS) of tissue smoke generated by the use of an electrosurgical instrument.

Patients recruited in the trial receive standard-of-care oral squamous cell carcinoma tumor excision surgery.

DETAILED DESCRIPTION:
Oral squamous cell carcinoma is the sixth common carcinoma and the cause of 1-2% of cancer related deaths in the world. The incidence of oral squamous cell carcinoma was 255 cases in Finland and 742 270 cases worldwide in year 2015. The number of cases per year has been increasing. The approximate age of tumor occurrence is usually between 60 - 70 years. The 5-year survival rate of all diagnosed oral squamous cell carcinoma cases in Finland during the years between 2014 and 2016 was 67% for women and 61% for men.

Early diagnostics is relevant, since oral squamous cell carcinoma tumors have a tendency to grow rapidly and metastasize early to regional lymphnodes and later on to lungs, liver and bones. Typical locations of the tumor are tongue, gums and sole of mouth.

The primary treatment option for oral squamous cell carcinoma is surgical removal of the tumor with 0,5 - 1cm healthy tissue margin. The aim of the operation is to remove the tumor entirely so that the healthy tissue margins are as sparing as possible and that the functional and cosmetic outcomes are as satisfactory as possible. Sufficient healthy tissue margin is one of the most important prognostic factors. Nevertheless, there is only little evidence based knowledge of sufficient healthy tissue margins.

Differential mobility spectrometry (DMS) based application called automatic tissue analysis (ATAS) can be utilized to identify tumor cells from healthy tissue. Tissue identification is done by analyzing tissue smoke that is generated by the use of an electrosurgical instrument called diathermy.

The objective of the trial is to test whether it is possible to identify oral squamous cell carcinoma tissue from normal oral mucosa by using ATAS. A 4mm punch biopsy of an oral squamous cell carcinoma tumor and a control biopsy of healthy oral mucosa will be collected from 30 - 40 patients undergoing oral tumor excision. The biopsies will be examined in the research laboratory with ATAS to test tissue recognition.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy diagnosed oral squamous cell carcinoma.
* Tumor diameter of 2 cm or larger.
* Operable patient that is willing to participate in the trial.

Exclusion Criteria:

* Tumor diameter less than 2 cm.
* Patient that is unwilling to take part in the trial.
* Patient that is not able to understand given information concerning the trial or to give concent to take part in the trial.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with oral squamous cell carcinoma and treated in the outpatient clinic of otorhinolaryngology in Tampere University Hospital, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of normal and cancerous tissue identification by differential mobility spectrometry | Through study completion, an average of 1 year
  The ATAS device records a molecular spectrum of the surgical smoke generated when the collected tissue samples are processed with an electrosurgical instrument in the research laboratory. The primary outcome of the study is to test the ability of the device to correctly distinguish cancerous tissue from normal tissue based on predicted differences in the spectrum.

SECONDARY OUTCOMES:
The influence of oral squamous cell carcinoma tumor thickness and infiltration depth on the resolution | Through study completion, an average of 1 year
  The overall thickness of the tumor and the infiltration depth of the tumor, both presented in millimetres, can have an effect on the resolution of cancerous tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Niku Oksala, M.D. Ph.D., Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
The research data will be published statistically and anonymously. A single participant can not be identified of the research data. Only the members of the research group will handle the individual participant data (IPD).

REFERENCES:
- [Background] P Economopoulou, A Psyrri. Epidemiology, risk factors and pathogenesis of squamous cell tumours. 2017 European Society for Medical Oncology (ESMO) Essentials for Clinicians and Neck Cancers Chapter 1
- [Background] Suusyöpä, Käypä Hoito -suositus 2019 (2019 Finnish Clinical Practice Guideline for Oral Carcinoma)
- [Background] McMahon J, O'Brien CJ, Pathak I, Hamill R, McNeil E, Hammersley N, Gardiner S, Junor E. Influence of condition of surgical margins on local recurrence and disease-specific survival in oral and oropharyngeal cancer. Br J Oral Maxillofac Surg. 2003 Aug;41(4):224-31. doi: 10.1016/s0266-4356(03)00119-0. PMID 12946663
- [Background] Anderson CR, Sisson K, Moncrieff M. A meta-analysis of margin size and local recurrence in oral squamous cell carcinoma. Oral Oncol. 2015 May;51(5):464-9. doi: 10.1016/j.oraloncology.2015.01.015. Epub 2015 Feb 21. PMID 25716108
- [Background] Sutton DN, Brown JS, Rogers SN, Vaughan ED, Woolgar JA. The prognostic implications of the surgical margin in oral squamous cell carcinoma. Int J Oral Maxillofac Surg. 2003 Feb;32(1):30-4. doi: 10.1054/ijom.2002.0313. PMID 12653229
- [Background] Lubek JE, Magliocca KR. Evaluation of the Bone Margin in Oral Squamous Cell Carcinoma. Oral Maxillofac Surg Clin North Am. 2017 Aug;29(3):281-292. doi: 10.1016/j.coms.2017.03.005. Epub 2017 May 24. PMID 28551338
- [Background] Covington JA, van der Schee MP, Edge AS, Boyle B, Savage RS, Arasaradnam RP. The application of FAIMS gas analysis in medical diagnostics. Analyst. 2015 Oct 21;140(20):6775-81. doi: 10.1039/c5an00868a. PMID 26205889
- [Background] Sutinen M, Kontunen A, Karjalainen M, Kiiski J, Hannus J, Tolonen T, Roine A, Oksala N. Identification of breast tumors from diathermy smoke by differential ion mobility spectrometry. Eur J Surg Oncol. 2019 Feb;45(2):141-146. doi: 10.1016/j.ejso.2018.09.005. Epub 2018 Oct 15. PMID 30366874
- See also: Citation 2: 2019 Finnish Clinical Practice Guideline for Oral Carcinoma — https://www.kaypahoito.fi/xmedia/khp/khp00032.pdf